CLINICAL TRIAL: NCT06258070
Title: Clinical Performance of Therapeutic Use of Botulinum Toxin in the Treatment of Bruxism: A Retrospective Study
Brief Title: Clinical Performance of Therapeutic Use of BTX for Bruxism
Acronym: BTX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Tahar Maamouri University Hospital (Other)
Responsible Party: Principal Investigator, Imen Turki Mehri, MD, Principal investigator, Mohamed Tahar Maamouri University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: University hospital Maamouri
Record Dates: First submitted 2024-01-20; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Myofascial Pain Syndrome; Myofascial Trigger Point Pain; Bruxism; Pain
Keywords: Botulinum toxin; treatment; bruxism; myofascial pain syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes; Bruxism; Pain | interventions — abobotulinumtoxinA; Botulinum Toxins

STUDY DESIGN:
Intervention Model Description: A retrospective cohort study of two samples of participants ( group with long-standing for more than one year, group with recent symptoms for less than one year), with a single-arm trial (all the participants had the same treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Duration of symptoms before BTX injections (Other): All the participants received BTX injections. Informed consent was obtained. Doses and sessions of injections varied between them according to the time of recurrence and the duration of the primary symptoms.
  The investigator carried out injections using Dysport (Ipsen Pharma, Germany). The toxin was reconstituted with 0.9% sodium chloride solution so that 0.1 ml corresponded to 25 U. The patient received the same doses in each session, delivered to TrPs detected by carefully palpating the muscle. 0.05 ml was injected into each TrPs.
  Interventions: Other: Abobotulinumtoxin A injection for bruxism

INTERVENTIONS:
Other: Abobotulinumtoxin A injection for bruxism — Trigger points were detected with careful palpating of the masticatory muscles (masseter and temporalis muscles) of patients suffering from bruxism. Each trigger point received 0,05 lm ol reconstituted solution of Abobotulinumtoxin A. Dysport (Ipsen Pharma, Germany) was reconstituted with 0.9% sodium chloride solution so that 0.1 ml corresponded to 25 U.
  Other Names: Botulinum toxin injection for bruxism

SUMMARY:
The goal of this clinical trial is to learn about the performance of botulinum toxin (BTX) injections for bruxism. Participants were divided into two groups according to the duration of the symptoms. The main question is whether BTX should be reserved for long-standing bruxism where the conventional methods failed or indicated as a first-line treatment. The investigator also compared the required doses and the frequency of treatment sessions between these two groups for a complete recovery.

DETAILED DESCRIPTION:
The effectiveness of botulinum toxin (BTX) in treating bruxism is recognized and well-established. This study aims to provide the most suitable condition for a better performance of BTX injections.

This retrospective study of a single-arm trial was conducted using a medical database of 67 patients who suffered from bruxism between 2009 and 2015, and who had total recovery after injection sessions. Patients were divided into two groups based on the duration of their bruxism. The main outcomes measured were: pain relief, the total number of injection sessions until total recovery, doses of BTX used, and recovery duration between two consecutive sessions. The treatment was stopped when bruxism disappeared.

The investigator carried out injections using Dysport (Ipsen Pharma, Germany). The toxin was reconstituted with 0.9% sodium chloride solution so that 0.1 ml corresponded to 25 U. The patient received the same doses in each session, delivered to trigger points (TrPs). 0.05 ml was injected into each TrP.

The level of statistical significance was set at p < 0,01. The Chi-square test and ANOVA table were used to compare differences according to injection sessions, doses of BTX, TrPs, and recovery duration between the two groups (with long-standing bruxism, and recent bruxism).

ELIGIBILITY:
Inclusion Criteria:

* Patients who self-reported having awake bruxism and recovered completely following BTX injections during the period ranging between 2009 and 2015. It includes patients who had previously occlusal splints and who should stop their use once the BTX injections were started.

Exclusion Criteria:

* Patients suffering from temporomandibular disorders or having a contraindication to BTX injection.

Ages: 37 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Correlation between doses of BTX and TrPs | 16 to 55 months
  The required doses of BTX were compared according to the number of trigger points found in both groups

SECONDARY OUTCOMES:
Comparison of the rate of injection sessions | 16 to 55 months
  The number of session of BTX injection for complete recovery was studied for both groups.
Correlation of the long standing symptoms and the time to recurrence | 16 to 55 months
  The time to recurrence was compared between individuals of both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Imen Mehri Turki, Dr, Principal Investigator — University hospital Mohamed Tahar Maamouri. Nabeul, Tunisia
Locations (1):
- Imen Mehri Turki, Nabeul, Tunisia

IPD SHARING:
Plan to Share IPD: No
If the study is published in a medical journal, data will be available for researchers.